CLINICAL TRIAL: NCT06101186
Title: The Effect of Nursing Counseling Based on Neuman Systems Model on Perceived Stress, Coping With Stress and Birth Outcomes Among Pregnant Women at High Risk of Pre-term Labor
Brief Title: The Effect of Nursing Counseling Perceived Stress, Coping and Birth Outcomes Among Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erzurum Technical University (Other)
Collaborators: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Ayşe Metin, Assistan Proffesor, Erzurum Technical University
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 040818
Record Dates: First submitted 2023-09-27; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Preterm Birth
Keywords: Risk of Preterm Labor; Neuman Systems Model; Stress; Coping with Stress; Birth Outcomes
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): Participants in the control group received standard nursing care provided by the institution where the research was conducted. After the study, we shared the materials developed for NPECP with the participants in the control group.
- Experimental group (Experimental): Nursing education and counseling practice to be applied to the experimental group was based on NSM. In the implementation of NPECP, the women were first met, and after the meeting, their informed consent was taken and they were included in the study. It was stated that the women in the experimental group were told that four scheduled interviews would be conducted online in a period of approximately 4 weeks. The women were given a telephone number where they could contact the researcher so that they could receive telephone/online counseling and were included in the whatsapp group with their permission.
  Interventions: Other: NPECP based on NSM

INTERVENTIONS:
Other: NPECP based on NSM — A comprehensive training booklet which integrated NPECP and NSM principles was sent to five experts for their evaluation and feedback. Among these experts, one was a physician who specialized in obstetrics and gynecology while the remaining individuals were nurses. Group training sessions were conducted online, with each group comprising 4-6 participants. These sessions spanned four weeks, with each session being held weekly and lasting for approximately 60-90 minutes. The training covered various topics - including pregnancy, pregnancy-related changes, pregnancy danger signs, premature birth, stress, stress symptoms, stress coping strategies, childbirth, the postpartum period and the challenges of parenting (particularly when dealing with a pre-term baby)
  Arms: Experimental group

SUMMARY:
Aim: The aim of this study is to determine the effect of the Pregnant Nursing Education and Counseling Program (HEGDAP), which is structured on the Neuman Systems Model, on the perception of stress, coping with stress and birth outcomes in pregnant women with preterm labor risk.

Method: This study was conducted with 60 pregnant women at risk of preterm labor, including 30 experimental and 30 control, non-randomized double-blind pregnant women using pretest, interim follow-up and posttest. Data were collected using a personal information form, Perceived Stress in Risky Pregnancies Questionnaire, Ways of Coping with Stress Scale and Birth Outcomes Evaluation Form. Nursing counseling based on Neuman's System Model was applied to the intervention group. Data were evaluated using analysis methods such as t-test, chi-square, etc.

DETAILED DESCRIPTION:
Although pregnancy is a physiological condition involving homeostatic adaptations, it is also a process that can subject pregnant women to stress and vulnerability. Pregnant women experience stress due to various factors such as bodily changes, hormonal fluctuations, physical symptoms, concerns about parenting, relationship issues, fear of childbirth, and the health of their baby. Risky pregnant women, compared to non-risky pregnant women, experience even more intense stress related to their own health and the health of their babies. The stressors faced by risky pregnant women include being diagnosed with a risky pregnancy, experiencing an unwanted pregnancy, encountering signs of danger during pregnancy, negative thoughts related to the baby, hospitalization, fear of childbirth, adolescent pregnancies, marital problems, lack of social support, economic concerns, and postpartum problems. Perceived stress during pregnancy can lead to negative birth outcomes such as preterm labor, spontaneous abortion, neonatal malformation, low birth weight, and prenatal developmental delay. Pregnant women reporting high stress have a 25% to 60% increased risk of preterm birth compared to those reporting low stress. A study found that pregnant women perceiving high stress during pregnancy were twice as likely to experience premature labor and twelve times more likely to give birth to a low birth weight baby. Another study showed that stressed pregnant women give birth an average of one and a half weeks earlier than healthy pregnant women. Stress is considered a modifiable factor that contributes to preterm birth, and eliminating its negative effects can help reduce the rate of preterm birth due to maternal stress.To cope with the stress associated with a risky pregnancy, it is crucial for pregnant women to utilize coping mechanisms they have used in the past and learn new coping strategies. However, 27.4 percent of pregnant women in Turkey feel that their ability to cope with stress is inadequate. It is recommended that nurses provide training and counseling to help pregnant women at risk of preterm birth cope with stress more effectively. Encouraging participation in stress-reduction programs that provide specific information, education, or relaxation methods is important for pregnant women at risk, and counseling should be provided toward the end of the second trimester. Nurses can contribute to better health outcomes for both the mother and the baby by supporting the use of appropriate stress-coping methods in high-risk pregnant women. In addition to addressing the individual information needs of nurses, systematic training and consultation on nutrition, rest, activity, sexual life, fetal growth and development, potential complications, and fetal movement monitoring should be provided to reduce the stress levels of pregnant women at risk of preterm birth. It is believed that structuring the training and counseling program based on nursing theory will enhance the benefits provided.

This research is conducted based on the nursing theorist Neuman's Systems Model (NSM), which focuses on concepts such as stress, coping with stress, and the environment. The Neuman Systems Model offers a holistic approach to care, going beyond the traditional concept of illness. It emphasizes interdisciplinary approaches to disease treatment, prevention, health education, and health promotion. No previous studies were found that monitored the results of providing training and counseling to pregnant women at risk of preterm birth using the Neuman Systems Model. This study aims to present an innovative approach to reducing perceived stress, improving stress coping, and supporting positive birth outcomes in pregnant women at risk of preterm labor by implementing the Pregnant Nursing Education and Counseling Program (PNECP) structured on the Neuman Systems Model.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* 24-28. Being in the gestational week (this interval was chosen because the risk of preterm birth is usually determined at the 24th week of pregnancy and fetuses born between 24-28 weeks have the chance to live in special environments)
* Ability to read and write in Turkish
* Ability to use a smart phone or computer
* Ability to continue online training
* Being pregnant with only one baby
* Ability to participate in trainings

Exclusion Criteria:

* Refusal to participate in the research
* Being unable to read and write Turkish and/or be a foreign national
* Difficulty in understanding and perceiving
* Inability to use a smartphone or computer
* Having a previous diagnosis of a psychiatric illness (the patient or physician states that he or she has previously been diagnosed with schizophrenia, bipolar disorder, anxiety disorder, or used medication for this reason) from a psychiatrist.
* Multiple pregnancy
* The gestational week is less than 24 weeks and more than 28 weeks
* Continuous hospitalization

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Risky Pregnancy Perceived Stress Question Form | 5 Minutes
  The Risky Pregnancy Perceived Stress Question Form (RPPS-QF) was developed by researchers to determine the stress perceived by pregnant women at high risk in the five life areas specified in the NSM. The RPPS-QF consists of a total of three dimensions and 35 items - comprised of the Physiological Domain (9 items), Psychological Domain (12 items) and Sociocultural-Developmental-Spiritual Domain (14 items). The Cronbach's alpha value of the form, prepared via a five-point Likert scale, is 0.86. The Cronbach's alpha value of the questionnaire was determined as 0.85 in the Psychological Domain, 0.67 in the Physiological Domain and 0.72 in the Sociocultural-Developmental-Spiritual Domain. As an individual's RPPS-QF score increases, it is held that their perceived stress increases.
Styles of Coping with Stress Scale | 5 minutes
  The Styles of Coping with Stress Scale (SCSS), as recorded via a 4-point Likert-type scale, was developed by Lazarus and Folkman.20 The Turkish validity of the 30-item form of the scale has been ascertained by Şahin and Durak.21 The Cronbach's alpha value of the scale was found to be 0.78. The scale covers the "seeking social support" (4 items), "optimistic" (5 items), "self-confident" (7 items), "helpless" (38 items) and "submissive" (6 items) approaches. The scale further consists of 5 sub-dimensions. Each item in the scale is assigned a score of between 0 and 3, whereby the scores for each factor are calculated separately. A higher score indicates that the person uses that style more.21 The Cronbach's alpha value of the scale in this study was determined as 0.89.
Birth Outcome Evaluation Form | 10 minutes
  The Birth Outcome Evaluation Form was developed by researchers to assess postpartum maternal and newborn outcomes.13,22-25 It includes questions, for each birth, as to its birth type, whether it was full-term or pre-term, the presence of any complications for both the mother and the baby, the Apgar scores at the 1st and 5th minutes and the location in which the mother and baby are monitored.
Pregnant women in the experimental group who applied the HEGDAP program, which was structured to the Neuman Systems Model, use more effective methods in coping with stress than before the program. | 1, minutes
  The Birth Outcome Evaluation Form was developed by researchers to assess postpartum maternal and newborn outcomes.13,22-25 It includes questions, for each birth, as to its birth type, whether it was full-term or pre-term, the presence of any complications for both the mother and the baby, the Apgar scores at the 1st and 5th minutes and the location in which the mother and baby are monitored.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Metin, Principal Investigator — Erzurum Technical University
Locations (1):
- Ayşe Metin, Yakutiye, Erzurum, Turkey (Türkiye)

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-12-27): https://cdn.clinicaltrials.gov/large-docs/86/NCT06101186/Prot_SAP_ICF_000.pdf